CLINICAL TRIAL: NCT06753149
Title: Clinical Application Research and Evaluation of Biomarkers Predicting Clopidogrel Resistance in Patients with Ischemic Stroke
Brief Title: Evaluation of the Efficacy of Novel Biomarkers in Predicting Clopidogrel Resistance in Patients with Ischemic Stroke
Status: Not yet recruiting | Type: Observational
Sponsor: Nanjing First Hospital, Nanjing Medical University (Other)
Responsible Party: Sponsor
Other Study IDs: KY20241217-06
Record Dates: First submitted 2024-12-23; First posted 2024-12-31 (Actual); Last update posted 2024-12-31 (Actual); Status verified 2024-12

CONDITIONS: Ischemic Stroke; TIA (Transient Ischemic Attack); Clopidogrel Resistance
MeSH Terms: conditions — Ischemic Stroke; Ischemic Attack, Transient

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole blood
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

GROUPS / COHORTS (2):
- Clopidogrel resistance: Definition of clopidogrel resistance (quantitative indicator): After patients take clopidogrel:
  1. The maximum platelet aggregation rate (%) value is greater than 50%;
  2. Compared before and after, clopidogrel inhibits platelet aggregation by less than 20%;
  3. The platelet aggregation inhibition of clopidogrel is 5 ohms or more (resistance method).
- Clopidogrel sensitivity

SUMMARY:
The goal of this observational study is to explore the potential efficacy of related biomakers in predicting clopidogrel resistance in patients with ischemic stroke. To be specific :

1. To investigate the relationship between the changes in ADP induced platelet aggregation rate, human plasma C4BPα concentration, mRNA expression levels of mARC1 and ABCC3-013 (splicing variant) in peripheral blood leukocytes, and the changes in the mRNA expression levels of ABCC3-013 (splicing variant) in selected hospitalized patients before and on the 3rd and 7th day after antiplatelet therapy, as well as on the 30th and 90th day after follow-up, in accordance with the current guidelines for secondary stroke prevention, and to explore the relative efficacy of each biomarker in predicting clopidogrel resistance;
2. To collect blood samples from patients, extract their DNA samples, perform CYP2C19 genotyping, validate and evaluate the predictive efficacy and clinical application value of a biomarker "panel" composed of multiple new and old biomarkers for predicting clopidogrel resistance.

ELIGIBILITY:
Inclusion Criteria:

* Age range: 18-80 years old. Within 72 hours after symptom onset (admission), the patient has started receiving "standard" antiplatelet therapy (which must include Plavix, taken alone or in combination)
* Diagnosed with mild, non cardiogenic, non disabling AIS (NIHSS score ≤ 3) or high-risk TIA (ABCD2 stroke risk assessment ≥ 4) based on the patient's symptoms, signs (such as hemiplegia, hemianopia, hemiparesis, aphasia, etc.) and various routine diagnoses and tests (including but not limited to neuroimaging, such as cranial CT, MRI, Doppler, etc.)

Exclusion Criteria:

* 72 hours after the onset of symptoms (admission), the patient began receiving "standard" antiplatelet therapy (including polivix, taken alone or in combination) for moderate or severe AIS (NIHSS score ≥ 5)
* Patients who require intravenous thrombolysis (using rt PA, urokinase, alteplase, or tiniprase, etc.)
* Mechanical intervention for thrombectomy
* Cardiogenic AIS (with concomitant atrial fibrillation)
* Embolic stroke of unknown origin (ESUS)
* Perioperative stroke
* Use anticoagulant drugs (such as warfarin, rivaroxaban, dabigatran etexils, etc.)
* Individuals with severe liver and kidney dysfunction
* Individuals allergic to clopidogrel or aspirin
* Individuals with a tendency towards bleeding (such as low platelet count or active gastric or intestinal ulcers)
* Individuals with a history of easy miscarriage or who are currently pregnant
* Patients with malignant tumors or life expectancy of less than 1 year

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: * Age range: 18-80 years old. Within 72 hours after symptom onset (admission), the patient has started receiving "standard" antiplatelet therapy (which must include Plavix, taken alone or in combination)
  * Diagnosed with mild, non cardiogenic, non disabling AIS (NIHSS score ≤ 3) or high-risk TIA (ABCD2 stroke risk assessment ≥ 4) based on the patient's symptoms, signs (such as hemiplegia, hemianopia, hemiparesis, aphasia, etc.) and various routine diagnoses and tests (including but not limited to neuroimaging, such as cranial CT, MRI, Doppler, etc.)
Sampling Method: Probability Sample
Enrollment: 800 (Estimated)
Dates: Start 2025-02-01 (Estimated); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Recurrent new stroke within 90 days after antiplatelet therapy (stroke recurrence) | From enrollment to the end of treatment at 90 days

IPD SHARING:
Plan to Share IPD: No